CLINICAL TRIAL: NCT00519766
Title: Assessment of Nicotine Metabolism Among Underserved Pregnant Women From NE SCRIPT
Brief Title: Examining a New Biomarker of Nicotine Use Among Pregnant Women Who Participated in the New England SCRIPT
Acronym: SCRIPT
Status: Completed | Type: Observational
Sponsor: Memorial Hospital of Rhode Island (Other)
Responsible Party: Principal Investigator, Donna R. Parker, Associate Professor of Family Medicine & Epidemiology, Memorial Hospital of Rhode Island
Other Study IDs: 1392
Record Dates: First submitted 2007-08-21; First posted 2007-08-23 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Smoking; Tobacco Use Disorder
Keywords: Ratio of 3-Hydroxycotinine to Cotinine; Nicotine Metabolism; Pregnancy
MeSH Terms: conditions — Smoking; Tobacco Use Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Smoking during pregnancy is the single most preventable cause of illness and death among mothers and infants. Because of the stigma associated with tobacco use during pregnancy, pregnant women are less likely to disclose their smoking status to doctors or study researchers. This study will evaluate the use of a new biomarker of nicotine metabolism to estimate tobacco use in a group of pregnant women who participated in the New England Smoking Cessation and Reduction in Pregnancy Trial (SCRIPT).

DETAILED DESCRIPTION:
According to one source of 2004 data, approximately 13% of pregnant women reported smoking during the last 3 months of pregnancy. This is a major public health concern because smoking during pregnancy can lead to pregnancy complications and serious health problems in newborns, including a 50% increase in risk of low birth weight. The effect of tobacco exposure on infant birth weight may have long-term consequences, as fetal growth appears to be a predictor of coronary heart disease later in life. Pregnant women participating in clinical trials are less likely to disclose that they are smoking because of a desire to please study researchers. Therefore, a way to test for nicotine exposure is needed to accurately determine the number of pregnant women who smoke and the number of women who quit smoking during pregnancy.

A new biomarker of nicotine metabolism, the ratio of trans-3'-hydroxycotinine to cotinine (3-HC:C), may be an accurate estimate of nicotine exposure from tobacco. Trans-3'-hydroxycotinine and cotinine are both byproducts of nicotine that are excreted in the urine. The purpose of this study is to evaluate the effectiveness of the 3-HC:C ratio as a measure of prenatal tobacco smoke exposure between the first and third trimesters of pregnancy and to examine the use of the 3-HC:C ratio in relation to infant birth weight. In addition, changes in the 3-HC:C metabolism during pregnancy will be analyzed according to different racial and ethnic groups.

This study will enroll pregnant women who participated in the New England SCRIPT study, which drew from a predominately low-income, multi-ethnic population. There will be no study visits specifically for this study. Study researchers will analyze participants' SCRIPT study data from four surveys collected at baseline, during the third trimester, and 6 weeks and 6 months following childbirth. Researchers will analyze the following study data: smoking behavior, attitudes toward smoking, self-reported smoking status, number of cigarettes smoked per day, use of the assigned smoking cessation materials, and infant birth weight. Demographic information, including the participant's age, race and ethnicity, years of education, age of the fetus at study entry, and smoking practices of other household members, will also be examined. Urine samples collected from participants during the SCRIPT study will be analyzed for the 3-HC:C biomarker. This current study will use a new technique, liquid chromatography/atmospheric pressure ionization tandem spectrometry, to measure both cotinine and hydroxycotinine levels in the urine samples.

ELIGIBILITY:
Inclusion Criteria:

* Participated in the New England SCRIPT study

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 1997-09; Primary Completion 1999-03 (Actual); Study Completion 2002-11 (Actual)

PRIMARY OUTCOMES:
biochemically confirmed smoking quit rates

CONTACTS AND LOCATIONS:
Overall Officials: Donna R. Parker, ScD, Principal Investigator — Memorial Hospital of Rhode Island
Locations (1):
- Memorial Hospital of Rhode Island, Pawtucket, Rhode Island, United States

REFERENCES:
- [Result] Parker DR, Windsor RA, Roberts MB, Hecht J, Hardy NV, Strolla LO, Lasater TM. Feasibility, cost, and cost-effectiveness of a telephone-based motivational intervention for underserved pregnant smokers. Nicotine Tob Res. 2007 Oct;9(10):1043-51. doi: 10.1080/14622200701591617. PMID 17943620